CLINICAL TRIAL: NCT06868758
Title: Predictive Value of Tumor Vascular Normalization Scoring in the Response to Neoadjuvant Therapy in HER-2 Positive Breast Cancer: an Observational Study
Brief Title: Predictive Value of Tumor Vascular Normalization Scoring in HER-2 Positive Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Chongqing General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JRIIT-08-01
Record Dates: First submitted 2025-03-01; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HER2 Positive Breast Carcinoma; Neoadjuvant Therapy
Keywords: Tumor vascular normalization score; anti-HER2 antibody; Treatment efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Weeks
Biospecimen Retention: Samples With DNA — Blood samples & FFPE tumor blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HER2 positive breast cancer: Female breast cancer patients with histopathologically confirmed HER2-positive status (defined as HER2 immunohistochemistry [IHC] 3+ or HER2 IHC 2+ with positive confirmation by fluorescence in situ hybridization [FISH]) who are planned to receive neoadjuvant therapy, including chemotherapy and HER2-targeted regimens.

SUMMARY:
This study aims to evaluate the predictive value of the tumor vascular normalization score for the efficacy of neoadjuvant therapy in HER-2-positive breast cancer and explore its potential as a predictive biomarker. Through longitudinal observation of HER-2-positive breast cancer patients receiving standard treatment, we will analyze the correlation between vascular normalization scores and treatment responses (including objective response rate [ORR] and pathological complete response [pCR]) to optimize individualized therapeutic strategies. Additionally, an exploratory investigation will assess the impact of ginsenoside-containing formulations (e.g., Jinxing Capsule, Shenyi Capsule, Yiqi Jianpi Oral Liquid) on tumor vasculature and neoadjuvant therapy outcomes in HER-2-positive breast cancer, providing scientific insights for complementary therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients aged ≥18 years planned for neoadjuvant therapy.
* Histopathologically confirmed HER2-positive status (IHC 3+ or IHC 2+ with positive FISH confirmation).
* Mentally competent, no psychiatric disorders, with good compliance to treatment and follow-up.
* Voluntarily participate and provide written informed consent.

Exclusion Criteria:

* HER2-negative breast cancer.
* Pregnant, planning pregnancy, or lactating women.
* History of allergic predisposition or known/suspected allergy to study drugs.
* Participation in other clinical trials within the past 4 weeks or planned enrollment.
* Other conditions deemed ineligible by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female HER2 positive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between VNS and Therapeutic Outcomes | Patients will be assessed at the third week and fifth week after initiation of anti-HER2 therapy, as well as preoperatively (prior to surgery).
  Predictive value of VNI for pCR (ROC curve analysis). Unit of Measure: Statistical correlation coefficients (R²/AUC)

SECONDARY OUTCOMES:
Correlation between Ginsenoside Formulation Exposure and Tumor Vascular Normalization | Patients will be assessed at the third week and fifth week after initiation of anti-HER2 therapy, as well as preoperatively (prior to surgery).
  Ginsenoside Exposure Measurement:
  Tool: Plasma concentration via Ultra-Performance Liquid Chromatography-Tandem Mass Spectrometry (UPLC-MS/MS) Parameter: Total ginsenoside plasma concentration (unit: ng/mL) Time Frame: Pre-dose and at Cycle 3 Day 1 (C3D1) of neoadjuvant therapy
  Vascular Normalization Measurement:
  Tool: Dynamic Contrast-Enhanced MRI (DCE-MRI) with Extended Tofts Model Parameter: Vascular Normalization Index (VNI)
  Components:
  K<sup>trans</sup> (unit: min<sup>-1</sup>) Plasma volume fraction (v<sub>p</sub>, unit: %) Calculation: Composite score (range 0-1) derived from principal component analysis
  Statistical Correlation:
  Method: Spearman's rank correlation Unit: Spearman's ρ (range: -1 to 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing General Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided